CLINICAL TRIAL: NCT04034069
Title: Effects of Priming Intermittent Theta Burst Stimulation on Upper Limb Motor Recovery After Stroke: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Kenneth N. K. Fong, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSEARS20190718003
Record Dates: First submitted 2019-07-23; First posted 2019-07-26 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Stroke
Keywords: stroke; theta burst stimulation; upper limb; metaplasticity; priming
MeSH Terms: conditions — Stroke | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- cTBS + iTBS, in addition to robot-assisted training (Experimental): Participants will receive 10-session intervention of priming iTBS protocol (cTBS followed by iTBS, with an interval of 10 minutes). The stimulation will be delivered 3-5 sessions per week, lasting for 2-3 weeks. Participants will receive a 60-minute standard robot-assisted training after each stimulation session.
  Interventions: Device: Theta burst stimulation (TBS); Behavioral: Robot-assisted training
- Sham cTBS + iTBS, in addition to robot-assisted training (Active Comparator): Participants will receive 10-session intervention of non-primed, standard iTBS (sham cTBS followed by iTBS, with an interval of 10 minutes). The stimulation will be delivered 3-5 sessions per week, lasting for 2-3 weeks. Participants will receive a 60-minute standard robot-assisted training after each stimulation session.
  Interventions: Device: Theta burst stimulation (TBS); Behavioral: Robot-assisted training
- Sham cTBS + sham iTBS, in addition to robot-assisted training (Sham Comparator): Participants will receive 10-session intervention of sham stimulation (sham cTBS followed by sham iTBS, with an interval of 10 minutes). The stimulation will be delivered 3-5 sessions per week, lasting for 2-3 weeks. Participants will receive a 60-minute standard robot-assisted training after each stimulation session.
  Interventions: Device: Theta burst stimulation (TBS); Behavioral: Robot-assisted training

INTERVENTIONS:
Device: Theta burst stimulation (TBS) — Theta burst stimulation (TBS) is a potent form of repetitive transcranial magnetic stimulation (rTMS). Standard 600-pulse intermittent theta burst stimulation (iTBS) can enhance the corticomotor excitability, whereas standard 600-pulse continuous theta burst stimulation (cTBS) can suppress the corticomotor excitability. Sham stimulation uses an extreme low stimulation intensity which will not influence with corticomotor excitability. In the present study, real stimulation will be delivered in an intensity of 70% individual resting motor threshold while sham stimulation will be delivered in an intensity of 20% individual resting motor threshold.
  Other Names: Repetitive transcranial magnetic stimulation (rTMS)
Behavioral: Robot-assisted training — Fourier M2 upper limb rehabilitation robot (Fourier Intelligence Co. Ltd., Shanghai, China), will be used for upper limb proximal joints training. Fourier M2 upper limb rehab robot is an end-effector robot-assisted device. The device targets (1) flexion and extension of shoulder joint, (2) flexion and extension of elbow, (3) internal and external rotation of shoulder joint, and (4) abduction and adduction of shoulder joint, supported by tailored interactive TV games in the device. HandyRehab hand robot (Zunosaki Company Ltd., Hong Kong SAR) will be used for upper limb distal joints training. It is an exoskeleton over the hand which provides power-driven extension and grasping force to the fingers and thumb in order to assist the patient to open and close the paretic hand by means of surface electromyography-triggered from the signals through the forearm extensors and flexors.

SUMMARY:
The aim of this study is to investigate the effects of intermittent theta burst stimulation primed with continous theta burst stimulation (cTBS), on top of a standard robot-assisted training (RAT) on improving the upper limb motor functions of stroke survivors and to explore potential sensorimotor neuroplasticity with electroencephalography (EEG).

DETAILED DESCRIPTION:
Intermittent theta burst stimulation (iTBS) delivered to the affected primary motor cortex (M1) appears to enhance the brain response to rehabilitative intervention in patients with stroke. However, its clinical utility is highly affected by the response variability. New evidence has reported that preceding iTBS with a priming session of continuous theta burst stimulation (cTBS), may stabilize and even boost the facilitatory effect of iTBS on the stimulated M1, via metaplasticity. The aim of this study is to investigate the effects of iTBS primed with cTBS, on top of a standard robot-assisted training (RAT) on improving the upper limb motor functions of patients with chronic stroke and to explore potential sensorimotor neuroplasticity with electroencephalography (EEG). A three-arm randomized controlled trial (RCT) will be performed with an estimated total of 36 patients with subacute or chronic stroke. All participants will be randomly allocated to receive 10-session intervention of different TBS protocols (i.e., cTBS+iTBS, sham cTBS+iTBS and sham cTBS+sham iTBS), delivered for 3-5 sessions per week, lasting for 2-3 weeks. All participants will receive a 60-minute standard RAT after each stimulation session. Primary outcome will be Fugl-Meyer Assessment-Upper Extremity scores (FMA-UE). Secondary outcomes will be Action Research Arm Test (ARAT), kinematic outcomes generated during RAT as well as and EEG.

ELIGIBILITY:
Inclusion Criteria:

* with a diagnosis of a unilateral ischemic or hemorrhagic stroke;
* with stroke onset more than 6 months;
* from 18 to 75 years old;
* with mild to moderate impairment of upper limb functions due to stroke, measured using the Hong Kong Version of the Functional Test for the Hemiplegic Upper Extremity (FTHUE-HK) from level 2 to level 7;
* be able to understand verbal instruction and follow one-step commands;
* be able to give informed consent to participate;

Exclusion Criteria:

* any contraindications to rTMS/TBS, such as unstable medical condition, history of epileptic seizures, metal implants in vivo (eg, pacemaker, artificial cochlear, and implant brain stimulator), and a history of receiving craniotomy;
* previous diagnosis of any neurological disease excluding stroke;
* presence of any sign of cognitive problems (Abbreviated mental test Hong Kong version < 6/10);
* patients with extreme spasticity in any hemiplegic upper limb joint (Modified Ashworth score > 2) or severe pain that hinder the upper limb motor training;
* with other notable impairment of the upper limb affected by stroke, eg, recent fracture, severe osteoarthritis, congenital upper limb deformity
* any sign of anxiety or depression, as assessed by the Hospital Anxiety and Depression Scale.
* concurrent participation in an upper limb rehabilitation program or a medicine trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment-Upper Extremity scores (FMA-UE) | Baseline
  FMA-UE is a standard upper limb motor impairment assessment for stroke survivors. FMA-UE assesses voluntary movement, reflex activity, grasp and coordination.
Fugl-Meyer Assessment-Upper Extremity scores (FMA-UE) | 1 week
  FMA-UE is a standard upper limb motor impairment assessment for stroke survivors. FMA-UE assesses voluntary movement, reflex activity, grasp and coordination.
Fugl-Meyer Assessment-Upper Extremity scores (FMA-UE) | 2 weeks
  FMA-UE is a standard upper limb motor impairment assessment for stroke survivors. FMA-UE assesses voluntary movement, reflex activity, grasp and coordination.
Fugl-Meyer Assessment-Upper Extremity scores (FMA-UE) | 2 weeks after the completion of training
  FMA-UE is a standard upper limb motor impairment assessment for stroke survivors. FMA-UE assesses voluntary movement, reflex activity, grasp and coordination.
Action Research Arm Test (ARAT) | Baseline
  ARAT is a standard upper limb functional performance assessment for stroke survivors. ARAT assesses a patient's ability to handle objects differing in size, weight and shape. ARAT consists of 19 items grouped into four subscales: grasp, grip, pinch, and gross movement.
Action Research Arm Test (ARAT) | 1 week
  ARAT is a standard upper limb functional performance assessment for stroke survivors. ARAT assesses a patient's ability to handle objects differing in size, weight and shape. ARAT consists of 19 items grouped into four subscales: grasp, grip, pinch, and gross movement.
Action Research Arm Test (ARAT) | 2 week
  ARAT is a standard upper limb functional performance assessment for stroke survivors. ARAT assesses a patient's ability to handle objects differing in size, weight and shape. ARAT consists of 19 items grouped into four subscales: grasp, grip, pinch, and gross movement.
Action Research Arm Test (ARAT) | 2 weeks after the completion of training
  ARAT is a standard upper limb functional performance assessment for stroke survivors. ARAT assesses a patient's ability to handle objects differing in size, weight and shape. ARAT consists of 19 items grouped into four subscales: grasp, grip, pinch, and gross movement.

SECONDARY OUTCOMES:
Sensorimotor event-related desynchronization | Baseline
  Electroencephalographical assessment for cortical activation induced by movement and mirror visual feedback-based observation of movement
Sensorimotor event-related desynchronization | 2 weeks
  Electroencephalographical assessment for cortical activation induced by movement and mirror visual feedback-based observation of movement
Mean velocity | Baseline
  Mean velocity is a quantified assessment for movement efficiency during robot-assisted training with Fourier M2 device.
Mean velocity | 2 weeks
  Mean velocity is a quantified assessment for movement efficiency during robot-assisted training with Fourier M2 device.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Department of Rehabilitation Sciences, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
The data will be shared for research purpose upon reasonable request.

REFERENCES:
- [Derived] Zhang JJ, Bai Z, Fong KNK. Priming Intermittent Theta Burst Stimulation for Hemiparetic Upper Limb After Stroke: A Randomized Controlled Trial. Stroke. 2022 Jul;53(7):2171-2181. doi: 10.1161/STROKEAHA.121.037870. Epub 2022 Mar 23. PMID 35317611
- [Derived] Zhang JJ, Fong KNK. Effects of priming intermittent theta burst stimulation on upper limb motor recovery after stroke: study protocol for a proof-of-concept randomised controlled trial. BMJ Open. 2020 Mar 8;10(3):e035348. doi: 10.1136/bmjopen-2019-035348. PMID 32152174